CLINICAL TRIAL: NCT04727619
Title: Sleep Education for Elders Program Evaluation
Brief Title: Evaluation of SLEEP Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Robin Tucker, Assistant Professor, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00003748
Record Dates: First submitted 2020-10-20; First posted 2021-01-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analyses will be done by blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants who participated in the SLEEP program.
  Interventions: Behavioral: SLEEP program
- Control (No Intervention): Participants who did not participate in the SLEEP program.

INTERVENTIONS:
Behavioral: SLEEP program — SLEEP is a 6-week educational program designed to improve sleep hygiene and habits.
  Arms: Experimental

SUMMARY:
This study tests the effectiveness of a new educational intervention designed to improve sleep outcomes among an older adult population.

ELIGIBILITY:
Inclusion Criteria:

* participants who choose to enroll in the SLEEP program

Exclusion Criteria:

* younger than 40 years of age

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sleep quality: Pittsburgh Sleep Quality Index | immediately after the program
  Change in sleep quality as measured by Pittsburgh Sleep Quality Index. Scores range from 0-21 with higher scores representing worse outcomes.
Sleep quality: Pittsburgh Sleep Quality Index | Six months after program completion
  Change in sleep quality as measured by Pittsburgh Sleep Quality Index. Scores range from 0-21 with higher scores representing worse outcomes.
Sleep duration | immediately after the program
  Change in sleep duration (hours and minutes) as measured by Pittsburgh Sleep Quality Index
Sleep duration | Six months after program completion
  Change in sleep duration (hours and minutes) as measured by Pittsburgh Sleep Quality Index
Daytime sleepiness | immediately after the program
  Change in daytime sleepiness measured by Epworth Sleepiness Scale. Scale scoring ranges from 0-24, with higher scores indicating worse outcomes.
Daytime sleepiness | Six months after program completion
  Change in daytime sleepiness measured by Epworth Sleepiness Scale. Scale scoring ranges from 0-24, with higher scores indicating worse outcomes.
Insomnia symptoms | immediately after the program and six months later
  As measured by Insomnia Severity Index. Scores range from 0-28 with higher scores indicating worse outcomes.
Insomnia symptoms | Six months after program completion
  As measured by Insomnia Severity Index. Scores range from 0-28 with higher scores indicating worse outcomes.
Sleep hygiene habits | immediately after the program
  As measured by Sleep Hygiene Index. Scores range from 0-52 with higher scores indicating worse outcomes.
Sleep hygiene habits | Six months after program completion
  As measured by Sleep Hygiene Index. Scores range from 0-52 with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Sleep-related knowledge | immediately after the program
  As measured by several questions related to sleep health and hygiene
Sleep-related knowledge | six months later
  As measured by several questions related to sleep health and hygiene
Sleep satisfaction: questions measuring personal satisfaction with sleep quality and duration | immediately after the program
  As measured by questions measuring personal satisfaction with sleep quality and duration
Sleep satisfaction: questions measuring personal satisfaction with sleep quality and duration | six months later
  As measured by questions measuring personal satisfaction with sleep quality and duration
Program satisfaction: questions and comments related to program experiences | immediately after the program
  As measured by questions and comments related to program experiences
Program satisfaction: questions and comments related to program experiences | six months later
  As measured by questions and comments related to program experiences

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States